CLINICAL TRIAL: NCT06165523
Title: Effect of Flavored Kefir Versus Flavored Milk on Time-Trial Performance in Endurance Master Athletes
Brief Title: Kefir Versus Milk on Time-Trial Performance in Masters Athletes
Acronym: KVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-23-71
Record Dates: First submitted 2023-11-16; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Gastrointestinal Complication; Exercise Performance; Aerobic Endurance
Keywords: Kefir; Milk; Aerobic Endurance; Exercise Performance; Gastrointestinal Symptoms
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomized, crossover.
Masking Description: Both participant and investigator are unmasked to treatment conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (Placebo Comparator): Water
  Interventions: Other: Water
- Flavored Kefir (Experimental): 1% Lowfat Kefir manufactured by Lifeway Kefir and containing 18 g of CHO, 10 g of protein, and 2 g of fat
  Interventions: Other: Flavored Kefir
- Flavored Milk (Active Comparator): 1% Lowfat Milk manufactured by Prairie Farms and containing 24 g of CHO, 8 g of protein, and 2.5 g of fat
  Interventions: Other: Flavored Milk

INTERVENTIONS:
Other: Water — 340 mL plain tap water consumed immediately following glycogen depleting exercise
  Arms: Water
Other: Flavored Kefir — 320 mL kefir consumed immediately following glycogen depleting exercise
  Arms: Flavored Kefir
Other: Flavored Milk — 240 mL flavored milk consumed immediately following glycogen depleting exercise
  Arms: Flavored Milk

SUMMARY:
The purpose of this study is to determine the effects of added probiotic cultures to a carbohydrate + protein recovery beverage compared to a similar recovery beverage without probiotic cultures, in its ability to impact endurance performance, perceived ratings of gastrointestinal symptoms and markers of inflammation and intestinal damage.

DETAILED DESCRIPTION:
In a randomized, crossover fashion, the investigators will assess changes in exercise performance, gastrointestinal symptom rating scale scores, as well as interleukin-6 and intestinal fatty-acid binding protein levels following consumption of either water, kefir or flavored milk.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Normotensive (seated, resting systolic blood pressure < 140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (< 90 beats per minute).
* Age between 40 and 75 years of age
* Body Mass Index <30 kg/m2 or Body Fat <30% for females and <25% for males
* Performing aerobic exercise > 150 mins/week and training for at least 3 years
* Well-trained will be defined as athletes that meet two of the four following criteria: training frequency is 3-7 sessions/week; duration of training sessions is 60-240 min; training background is at least 3 y; race frequency is at least once a year.

Exclusion Criteria:

* Individuals currently diagnosed or being treated for any cardiac, respiratory, endocrine, psychiatric, musculoskeletal, renal, hepatic, neuromuscular or metabolic disease or disorder that in the judgement of the study participant's personal physician or research nurse that will preclude their safe participation or will contraindicate quality control over the collected data
* Individuals currently diagnosed with or are being treated for celiac disease, lactose intolerance, digestive insufficiencies or other gastrointestinal complications such as irritable bowel syndrome, ulcerative colitis, etc.

Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence.

* Smokers or individuals who have quit smoking within the last 6 months
* Participants that are unwilling to refrain from caffeine, nicotine, and alcohol intake for 12 hours prior to each study visit.
* Known sensitivity to any ingredient in the test formulations as listed in the Nutrition Facts label.
* Individuals who are determined to be on a ketogenic diet.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Participants that are unwilling to refrain from taking biotin at a minimum of 72 hours before visit 3 through the end of the study due to potential interference with laboratory analyses.
* Individuals taking a medication known to impact digestive function or hormonal functions that may impact how our body digests, absorbs or metabolizes nutrients
* Individuals that are currently taking a probiotic or a dietary supplement that may impact digestive function or hormonal function that may impact how our body digests, absorbs or metabolizes nutrients
* Participants that are unwilling to refrain from fermented foods and yogurt, as well as maintain normal consumption levels of prebiotics throughout the study.
* Pregnant women, women trying to become pregnant, or nursing women.
* Individuals who indicate they are actively restricting calories or attempting to lose weight.
* Participants that are unwilling to keep their self-directed training protocols the same throughout the course of the study
* Participants that are unwilling to wear the same shoes and similar clothing for all testing visits.
* Individuals who participate in aerobic exercise < 2 days/week or have been aerobically training < 3 years
* Individuals that do not meet the criteria to be defined as well-trained
* Unwillingness to intake a supplement or follow the study protocol
* Any other condition which in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose a significant risk to the subject.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Aerobic Performance Times | Through study completion, an average of 3 weeks
  5 kilometer running time-trial on a curved, non-motorized treadmill

SECONDARY OUTCOMES:
Blood Interleukin-6 | Through study completion, an average of 3 weeks
  Blood interleukin-6 concentrations in response to intense exercise
Blood Intestinal fatty-acid binding protein | Through study completion, an average of 3 weeks
  Blood Intestinal fatty-acid binding protein concentrations in response to intense exercise
Gastrointestinal Symptoms | Through study completion, an average of 3 weeks
  Gastrointestinal Symptoms measured using the Gastrointestinal Symptoms Rating Scale (GSRS) in response to intense exercise. The scale asks 15 questions, and asks participants to rate their gastrointestinal symptoms on a 7 point scale with 0 being no discomfort at all and 7 being very severe discomfort. Lower total GSRS scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make IPD available to other researchers